CLINICAL TRIAL: NCT02074657
Title: "LANK-2": Activated and Expanded NK Cell Immunotherapy Together With Salvage Chemotherapy in Children, Adolescents and Young Adults With Relapsed or Refractary Acute Leukemia
Acronym: LYDIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Antonio Pérez Martínez, MD, Servicio de Hemato-Oncología Pediátrica, Hospital Universitario La Paz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-005146-38
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Relapsed/Refractory Paediatric Acute Leukaemia
Keywords: Immunotherapy; NKAEs; Expanded haploidentical natural killer cells; Activated natural killer cells
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Activated natural killer cells (Experimental)
  Interventions: Biological: Activated and expanded natural killer cells (NKAEs)

INTERVENTIONS:
Biological: Activated and expanded natural killer cells (NKAEs) — Activated and expanded natural killer cells (NKAEs) from haploidentical donor

SUMMARY:
To determine safety profile of immunotherapy with natural killer cells and activated expanded (NKAEs) after salvage chemotherapy in children, adolescents and young adults with relapsed or refractary acute leukemia

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 0 and 23 years of age with diagnosis of acute lymphoblastic leukemia, in second relapse situation, posttransplant relapse or refractary, or
2. Patients between 0 and 23 years of age with diagnosis of acute myeloblastic leukemia, relapsed or refractary. (Patient must meet inclusion criteria 1 or 2)
3. Lansky index > 60%
4. Mild (<2) functional organs alteration (hepatic, renal, respiratory) according to National Cancer Institute criteria (NCI CTCAE v4).
5. Left ventricular ejection fraction > 39%
6. To grant informed consent in accordance with the current legal regulations.
7. Presence of a compatible haploidentical donor (father or mother or brother).

Exclusion Criteria:

1. Patients with history of bad therapeutical compliance
2. Patients not valid after psycho-social evaluation
3. Positive HIV serology

Max Age: 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2014-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
To assess the safety of activated and expanded NK cell (NKAE) immunotherapy after salvage chemotherapy in patients with relapsed or refractary acute leukemia | 2 months after infusion
  Number of patients with adverse events according to NCI-CTCAE v4.0 CRITERIA as a measure of safety and tolerability

SECONDARY OUTCOMES:
Incidence of episodes of febrile neutropenia, bacteriemia or viral or fungal infections | End of infusion and follow-up (2 months and 1 year)
Days of hematological recovery (neutrophils >500/microL, lymphocytes >250/microL and platelets >50.000/microL), days of hospitalization, in each cycle Immune | End of infusion and follow-up (2 months and 1 year)
Objective response rate according to cytomorphic and by "minimal residual disease" criteria (cytometry and/or real time PCR) at the end of the treatment | End of infusion and follow-up (2 months and 1 year)
Immune reconstitution: Median of T-cell , B, NK, Natural Killer T cell (NKT) and dendritic cells count and subpopulations of T and NK lymphocytes (cel/microL) during posttreatment follow-up period. | End of infusion and follow-up (2 months and 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pérez-Martínez, MD, PhD, Study Chair — Hospital Infantil Universitario La Paz
Locations (2):
- Spain (2):
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Infantil Universitario La Paz, Madrid, Madrid

REFERENCES:
- [Derived] Vela M, Corral D, Carrasco P, Fernandez L, Valentin J, Gonzalez B, Escudero A, Balas A, de Paz R, Torres J, Leivas A, Martinez-Lopez J, Perez-Martinez A. Haploidentical IL-15/41BBL activated and expanded natural killer cell infusion therapy after salvage chemotherapy in children with relapsed and refractory leukemia. Cancer Lett. 2018 May 28;422:107-117. doi: 10.1016/j.canlet.2018.02.033. Epub 2018 Feb 23. PMID 29477379